CLINICAL TRIAL: NCT01069939
Title: A Phase III Multinational, Multicenter, Randomized, Double-blind, Parallel-group, Comparative Efficacy and Safety Study of D961H (20 mg Once Daily) Versus Placebo for Prevention of Gastric and/or Duodenal Ulcers Associated With Continuous Low-dose Aspirin (LDA) Use
Brief Title: Comparative Efficacy & Safety Study of D961H Versus Placebo for the Prevention of Gastric and Duodenal Ulcers With Low-dose Aspirin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D961PC00001
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-10

CONDITIONS: Prevention
Keywords: Gastric ulcer; Duodenal ulcer; Low-dose aspirin
MeSH Terms: conditions — Stomach Ulcer; Duodenal Ulcer | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esomeprazole 20mg (Experimental): Esomeprazole 20mg once daily oral
  Interventions: Drug: Esomeprazole
- Placebo (Placebo Comparator): Placebo once daily oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — 20mg, capsule, 72 weeks
  Arms: Esomeprazole 20mg
Drug: Placebo — Placebo, capsule, 72 weeks
  Arms: Placebo

SUMMARY:
To assess the efficacy of D961H 20 mg once daily (q.d.) versus placebo in continuous treatment involving patients with a history of gastric and/or duodenal ulcers receiving daily Low-dose aspirin therapy by evaluating time from randomisation to occurrence of gastric and/or duodenal ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent before starting the study-related procedures and examinations
* Patients who have the history of gastric and/or duodenal ulcer.
* A diagnosis of a chronic condition (angina pectoris, myocardial infarction and ischemic cerebrovascular disorder, etc., requiring prevention of thrombosis or embolism) which requires taking the prescribed LDA during the study treatment period.

Exclusion Criteria:

* Having gastric or duodenal ulcer (except for ulcer scar).
* History of esophageal, gastric or duodenal surgery, except for simple closure of perforation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kentaro Sugano, MD, PhD, Principal Investigator — Jichi Medical University
Locations (46):
- Japan (36):
  - Research Site, Yotsukaidou, Chiba
  - Research Site, Fukui-shi, Fukui
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu-Shi, Fukuoka
  - Research Site, Onga-Gun, Fukuoka
  - Research Site, Yukuhashi, Fukuoka
  - Research Site, Fukushima, Fukushima
  - Research Site, Kōriyama, Fukushima
  - Research Site, Nihommatsu, Fukushima
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Kure, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Amagasaki, Hyōgo
  - Research Site, Itami, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Nishinomiya, Hyōgo
  - Research Site, Higashi-ibaraki,, Ibaraki
  - Research Site, Komatsu, Ishikawa-ken
  - Research Site, Nomi, Ishikawa-ken
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Uji, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Daitō, Osaka
  - Research Site, Kishiwada, Osaka
  - Research Site, Matsubara, Osaka
  - Research Site, Minato, Osaka
  - Research Site, Yao, Osaka
  - Research Site, Hanyū, Saitama
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Shimotsuke, Tochigi
  - Research Site, Chūō, Tokyo
  - Research Site, Minato, Tokyo
  - Research Site, Shinagawa, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Shimonoseki, Yamaguchi
- South Korea (5):
  - Research Site, Gangneung, Gangwon-do
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Seoul
- Taiwan (5):
  - Research Site, Niao-Song-Shiang, Kaohsiung
  - Research Site, Kweishan Shiang, Taoyuan Hsien
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei

REFERENCES:
- [Derived] Sugano K, Choi MG, Lin JT, Goto S, Okada Y, Kinoshita Y, Miwa H, Chiang CE, Chiba T, Hori M, Fukushima Y, Kim HS, Chang CY, Date M; LAVENDER Study Group. Multinational, double-blind, randomised, placebo-controlled, prospective study of esomeprazole in the prevention of recurrent peptic ulcer in low-dose acetylsalicylic acid users: the LAVENDER study. Gut. 2014 Jul;63(7):1061-8. doi: 10.1136/gutjnl-2013-304722. Epub 2013 Dec 10. PMID 24326741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled on 4 February 2010. On 20 May 2011, the efficacy analysis was completed based on positive results of an interim analysis so that the efficacy data in this report are at the interim analysis. To evaluate the safety, the study was continued. The last participant completed the study on 9 November 2011.
Pre-assignment Details: Out of 914 enrolled participants, 430 participants were assigned , but 484 participants were not assigned. The major reasons of no assignment were 'Did not meet eligibility criteria' (462 participants) and 'Voluntary discontinuation by participant' (21 participants). After 366 participants were randomised, the interim analysis was done.
Period: Randomised and Included in the Analyses
Arm/Group | Esomeprazole 20mg | Placebo
Started | 213 | 214
Completed | 164 | 137
Not Completed | 49 | 77
Not completed — Adverse Event | 17 | 22
Not completed — Withdrawal by Subject | 15 | 12
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Study-specific withdrawal criteria | 7 | 33
Not completed — Eligibility criteria not fulfilled | 4 | 3
Not completed — Use of prohibited concomitant drug | 4 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Removal | 1 | 0
Period: At Data Cut Off Date (26 Feb 2011)
Arm/Group | Esomeprazole 20mg | Placebo
Started | 213 | 214
Completed | 182 | 182
Not Completed | 31 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 20mg | Placebo | Total
Number analyzed (Participants) | 213 | 214 | 427
Age, Customized [Number; unit: Participants]
  <=64years | 85 | 71 | 156
  Between 65 and 74 years | 82 | 89 | 171
  >=75 years | 46 | 54 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 46 | 89
  Male | 170 | 168 | 338
Region of Enrollment [Number; unit: Participants]
  Taiwan | 22 | 21 | 43
  Japan | 160 | 160 | 320
  Korea, Republic of | 31 | 33 | 64
Helicobacter pylori status [Number; unit: Participants] — 8 participants had a missing for this measurement (3 participants in Esomeprazole 20 mg group and 5 participants in Placebo group). Negative means a patient had no Helicobacter pylori infection and Positive means a patient had Helicobacter pylori infection.
  Participants
    Positive | 93 | 93 | 186
    Negative | 117 | 116 | 233

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Occurrence of Gastric and/or Duodenal Ulcers up to Data Cut-off Date for Interim Analysis.
Description: Assessments for occurrence of gastric and/or duodenal ulcers were performed every 12 weeks after randomisation. The numbers of participants with recurrence of gastric and/or duodeal ulcers were analysed every 12 weeks up to 48 weeks.
Time Frame: From randomisation to up to 48 weeks (Maximum follow-up period at the interim analysis)
Population: Participants not taking investigational drug were not included. In total 364 participants were included in the efficacy evaluation at the interim analysis. 24 of the 364 total participants had an occurrence of gastric and/or duodenal ulcers by the 48-week assessment.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 182 | 182
Participants
  0 - 12 weeks | 1 | 16
  13 - 24 weeks | 1 | 4
  25 - 36 weeks | 0 | 2
  37 - 48 weeks | 0 | 0
Statistical Analysis 1: Comparison: Esomeprazole 20mg vs Placebo; The above two groups were compared; Test type: Superiority or Other; p < 0.001, Log Rank — An interim analysis was done so that the significance level was adjusted using the Pocock-like alpha-spending function with Lan-DeMets approach. The adjusted significance level was the two-sided 3.35%; Hazard Ratio (HR) = 0.09, 96.65% CI 2-sided [0.02 to 0.41]

2. Secondary Outcome: Change in Degree of Gastric Mucosal Lesion by Modified Lanza Scale From Baseline to Last Measurement up to Week 48
Description: Modified Lanza scale attributes the degree of gastric mucosal lesion, graded on a 5 point scale (0=No hemorrhage, no erosion, 1=One hemorrhage or one erosions, 2=2-10 hemorrhages or erosions, 3=11-25 hemorrhages or erosions, 4=More than 25 hemorrhages or erosions, or ulcer). Higher scores indicate greater severity of gastric mucosal lesion.
Time Frame: Up to 48 weeks (Baseline to last measurement)
Population: Participants who had LANZA scores at both baseline and post-dose were included into this analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 144 | 145
Scores on a scale | -0.4 (0.6) | 1.3 (1.6)

3. Secondary Outcome: Number of Participants With Reflux Esophagitis Evaluated by the LA Classification up to Week 48.
Description: Endoscopy was conducted at 12, 24, 36 and 48 weeks after randomisation. At the endoscopy, participants was evaluated whether they have reflux esophagitis or not.
Time Frame: 12, 24, 36 and 48 weeks
Population: Patients with endoscopy were included in the analyses at 12, 24, 36 and 48 weeks after randomisation.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 141 | 138
Participants
  12 weeks | 0 | 9
  24 weeks | 1 | 6
  36 weeks | 0 | 3
  48 weeks | 0 | 0

4. Secondary Outcome: Change in the Severity of Epigastric Pain From Baseline to Last Measurement up to Week 48
Description: The severity of epigastric pain at baseline and the last measurement up to 48 weeks was obtained (None, Mild, Moderate, Severe). If the value at the last was better in a participant, the participant was categorized into "Improved". If the value was same, categorised into "Unchanged". If the value was worsened, categorise into "Worsened".
Time Frame: Up to 48 weeks (Baseline to last measurement)
Population: Participants who had the measurements of epigastric pain at baseline and post-dose up to 48 weeks were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 168 | 172
Participants
  Improved | 11 | 16
  Unchanged | 153 | 145
  Worsened | 4 | 11

5. Secondary Outcome: Change in the Severity of Heartburn From Baseline to Last Measurement up to Week 48.
Description: The severity of heartburn at baseline and the last measurement up to 48 weeks was obtained (None, Mild, Moderate, Severe). If the value at the last was better in a participant, the participant was categorized into "Improved". If the value was same, categorised into "Unchanged". If the value was worsened, categorise into "Worsened".
Time Frame: Up to 48 weeks (Baseline to last measurement)
Population: Participants who had the measurements of heartburn at baseline and post-dose up to 48 weeks were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 168 | 172
Participants
  Improved | 7 | 6
  Unchanged | 158 | 154
  Worsened | 3 | 12

6. Secondary Outcome: Change in the Severity of Anorexia From Baseline to Last Measurement up to Week 48
Description: The severity of anorexia at baseline and the last measurement up to 48 weeks was obtained (None, Mild, Moderate, Severe). If the value at the last was better in a participant, the participant was categorized into "Improved". If the value was same, categorised into "Unchanged". If the value was worsened, categorise into "Worsened".
Time Frame: Up to 48 weeks (Baseline to last measurement)
Population: Participants who had the measurements of anorexia at baseline and post-dose up to 48 weeks were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 168 | 172
Participants
  Improved | 9 | 10
  Unchanged | 156 | 153
  Worsened | 3 | 9

7. Secondary Outcome: Change in the Severity of Abdomen Enlarged Feeling From Baseline to Last Measurement up to Week
Description: The severity of abdomen enlarged feeling at baseline and the last measurement up to 48 weeks was obtained (None, Mild, Moderate, Severe). If the value at the last was better in a participant, the participant was categorized into "Improved". If the value was same, categorised into "Unchanged". If the value was worsened, categorise into "Worsened".
Time Frame: Up to 48 weeks (Baseline to last measurement)
Population: Participants who had the measurements of abdomen enlarged feeling at baseline and post-dose up to 48 weeks were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 168 | 172
Participants
  Improved | 18 | 24
  Unchanged | 141 | 141
  Worsened | 9 | 7

8. Secondary Outcome: Change in the Severity of Nausea and/or Vomiting From Baseline to Last Measurement up to Week 48
Description: The severity of Nausea and/or Vomiting at baseline and the last measurement up to 48 weeks was obtained (None, Mild, Moderate, Severe). If the value at the last was better in a participant, the participant was categorized into "Improved". If the value was same, categorised into "Unchanged". If the value was worsened, categorise into "Worsened".
Time Frame: Up to 48 weeks (Baseline to last measurement)
Population: Participants who had the measurements of Nausea and/or Vomiting at baseline and post-dose up to 48 weeks were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 168 | 172
Participants
  Improved | 8 | 5
  Unchanged | 160 | 154
  Worsened | 0 | 13

9. Secondary Outcome: Change in the Severity of Discomfort in the Stomach From Baseline to Last Measurement up to Week 48
Description: The severity of Discomfort in the stomach at baseline and the last measurement up to 48 weeks was obtained (None, Mild, Moderate, Severe). If the value at the last was better in a participant, the participant was categorized into "Improved". If the value was same, categorised into "Unchanged". If the value was worsened, categorise into "Worsened".
Time Frame: Up to 48 weeks (Baseline to last measurement)
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 168 | 172
Participants
  Improved | 13 | 15
  Unchanged | 150 | 148
  Worsened | 5 | 9

10. Secondary Outcome: Number of Participants With Adverse Events
Description: Participants who had at least adverse events (AE) which occurred after receiving study drug were counted.
Time Frame: Up to 70 weeks at the longest
Population: All participants who received any study drug were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20mg | Placebo
Number analyzed (Participants) | 214 | 213
Participants
  Adverse event | 155 | 139
  Adverse event (Frequency>=5%) | 70 | 53
  Death | 0 | 0
  Serious adverse event other than death | 17 | 15
  Adverse event leading to discontinuation of study | 17 | 22
  Drug-related adverse event | 31 | 29
  Severe adverse event | 7 | 10

ADVERSE EVENTS:
Arm/Group | Esomeprazole 20mg | Placebo
Serious Adverse Events (participants affected / at risk) | 17/214 | 15/213
Other Adverse Events (participants affected / at risk) | 70/214 | 53/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20mg (N=214) | Placebo (N=213)
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Renal Infarct (Renal and urinary disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostatic Specific Antigen Increased (Investigations) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 1 | 0
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Cholangitis Acute (Hepatobiliary disorders) | 1 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 1
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Cardiac Myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0
Brain Stem Haemorrhage (Nervous system disorders) | 2 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 2
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20mg (N=214) | Placebo (N=213)
Duodenitis (Gastrointestinal disorders) | 4 | 11
Gastric Polyps (Gastrointestinal disorders) | 11 | 1
Constipation (Gastrointestinal disorders) | 12 | 11
Nasopharyngitis (Infections and infestations) | 43 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs were prohibited to disclose all information related to this study without AZ approval before this study was completed.